CLINICAL TRIAL: NCT00590590
Title: Safety and Efficacy of Two Vaginal Products Versus Placebo in Patients With Vaginal Discomfort
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDC-201-601-669020
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Lidocaine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 3 (Placebo) (Placebo Comparator)
  Interventions: Drug: placebo
- 1 (Lidocaine) (Experimental)
  Interventions: Drug: lidocaine
- 2 (Lidocaine/Diphenhydramine) (Experimental)
  Interventions: Drug: Lidocaine/Diphenhydramine

INTERVENTIONS:
Drug: Lidocaine/Diphenhydramine — semi solid, twice weekly, 4 months
  Arms: 2 (Lidocaine/Diphenhydramine)
Drug: lidocaine — semi solid, twice weekly for 4 months
  Arms: 1 (Lidocaine)
Drug: placebo — semi solid, twice weekly for 4 months
  Arms: 3 (Placebo)

SUMMARY:
This study will evaluate the efficacy and safety of two vaginal products compared with that of placebo to determine if the two products are better than placebo in the relief of vaginal discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have sought doctor's care for this condition.
* Patients must be having menstrual cycles.

Exclusion Criteria:

* Patients must not have any vaginal infections.
* Patients must not be pregnant or nursing.
* Must not be receiving any other medicinal therapies or any medications that would interfere with the outcome of the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Lumara Health, Inc.
Locations (48):
- United States (41):
  - Montgomery Women's Health Associates, P.C., Montgomery, Alabama
  - Star W. Research, Chandler, Arizona
  - Precision Trials LLC, Phoenix, Arizona
  - Searcy Medical Center, Searcy, Arkansas
  - Universal Biopharma Research Institute, Inc., Dinuba, California
  - San Diego Clinical Research Center, San Diego, California
  - Red Rocks OB/GYN, Lakewood, Colorado
  - Taylor Associates/Gynecology, Farmington, Connecticut
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Clinical Research of Tampa Bay, Hudson, Florida
  - Innovative Research of W. Florida, Largo, Florida
  - Women's Health Care Specialists, PC, Paw Paw, Florida
  - Tampa Bay Women's Healthcare Alliance, LLP, Tampa, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Atlanta Women's Research Institute, Inc., Atlanta, Georgia
  - Atlanta North Gynecology, PC, Roswell, Georgia
  - Womans Clinic, Boise, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Women's Health Practice, LLC, Champaign, Illinois
  - Northern Indiana Womens Health Research, South Bend, Indiana
  - Female Pelvic Medicine and Urogynecology, Grand Rapids, Michigan
  - Boro Park ObGyn, Brooklyn, New York
  - Eastern Carolina Womens Center, New Bern, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Winston-Salem Woman Care, PA, Winston-Salem, North Carolina
  - Holzer Clinic, Gallipolis, Ohio
  - HWC Women's Research Center, Miamisburg, Ohio
  - Advanced Clinical Research, Medford, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Advanced Clinical Concepts, West Reading, Pennsylvania
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Women's Care Center, PLC, Memphis, Tennessee
  - Gynecology and Obstetrics, P.C., Memphis, Tennessee
  - Professional Quality Research/Women Partners, Austin, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Woman's Hospital of Texas, Houston, Texas
  - Bexar Clinical Trials, Irving, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Salt Lake Women's Center, Sandy City, Utah
- Canada (7):
  - Gain Medical Centre, Coquitlam, British Columbia
  - Stephen Kaye, MD, North Vancouver, British Columbia
  - Southern Healthcare Centre, White Rock, British Columbia
  - Common Wealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - The Ottawa Hospital-Soundcare Medical Centre, Ottawa, Ontario
  - Royal Health Care Centre, Toronto, Ontario
  - Windsor Metropolitan Hospital, Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 31 physician offices in the US and Canada between 04Sep2007 to 18Mar2009.
Pre-assignment Details: Participants will undergo a screening period of two weeks prior to study assignment.
Groups:
- Lidocaine/Diphenhydramine (Combination): Lidocaine/Diphenhydramine (Combination) administered twice weekly for 4 months
- Lidocaine: Lidocaine administered twice weekly for 4 months
- Placebo: Placebo administered twice weekly for 4 months
Period: Overall Study
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Started | 39 | 39 | 27
Completed | 32 | 33 | 21
Not Completed | 7 | 6 | 6
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lost to Follow-up | 4 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Did not complete due to study closure | 1 | 1 | 1
Not completed — Did not complete study | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo | Total
Number analyzed (Participants) | 39 | 39 | 27 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 27 | 105
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (7.4) | 32 (9.0) | 32 (9.5) | 31 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 27 | 105
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 39 | 25 | 100
  Canada | 3 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Marinoff Dyspareunia Scale Score (MDSS) at End of Treatment (12 Weeks)
Description: The MDSS consists of a participant rating of their dyspareunia (painful sexual intercourse) on a 0- to 3-point scale. Each numerical value on the scale coincides with a level of pain experienced during sexual intercourse; 0 = no dyspareunia (no pain with intercourse) and 3 = completely prevents intercourse
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
scores on a scale | 1.8 (0.12) | 1.8 (0.12) | 1.7 (0.14)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = 0
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1

2. Secondary Outcome: Change From Baseline in Marinoff Dyspareunia Scale Score at End of Treatment (12 Weeks)
Description: 0-3 scale with 0=no dyspareunia and 3= completely prevents intercourse
Time Frame: Baseline -12 Weeks
Measure: Mean (Standard Error); unit: Score
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
Score | -0.6 (0.15) | -0.4 (0.13) | -0.7 (0.15)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3

3. Secondary Outcome: Change From Baseline in Overall Vulvar Vestibulitis Syndrome (VVS)-Related Discomfort Visual Analog Scale (VAS) Score at End of Treatment (12 Weeks) [0 = No Discomfort and 100 = Most Severe Discomfort]
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: Score
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
Score | -9.9 (3.48) | -3.8 (4.46) | -14.6 (4.56)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = -6.1
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 4.7
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 10.8

4. Secondary Outcome: Change From Baseline in Overall Intercourse-Related Pain Visual Analog Scale (VAS) Score at End of Treatment (12 Weeks) [0 = No Pain and 100 = Most Severe Pain]
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
Score | -10.3 (5.71) | -19.6 (4.42) | -19.3 (6.55)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = 9.3
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 9
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3

5. Secondary Outcome: Change From Baseline in Overall Vulvar Vestibulitis Symptoms Visual Analog Scale (VAS) Score at End of Treatment (12 Weeks) [0 = No Symptoms and 100 = As Bad as They Can be]
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: Score
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
Score | -10.4 (4.31) | -5.3 (4.47) | -16.3 (4.22)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = -5.1
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 5.9
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 11

6. Secondary Outcome: Change From Baseline in Tenderness (on a 0- to 3-point Scale) on Palpation at End of Treatment (12 Weeks) [Scale Rates the Severity of Pain; 0 =Absent and 3 = Severe]
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: Score
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 39 | 27
Score | -3.0 (0.70) | -1.7 (0.67) | -2.4 (0.75)
Statistical Analysis 1: Comparison: Lidocaine/Diphenhydramine (Combination) vs Lidocaine; Ha: Drug 1 < Drug 2; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3
Statistical Analysis 2: Comparison: Lidocaine/Diphenhydramine (Combination) vs Placebo; Ha: Drug 1 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6
Statistical Analysis 3: Comparison: Lidocaine vs Placebo; Ha: Drug 2 < Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.7

ADVERSE EVENTS:
Time Frame: 16 weeks for each subject
Description: Adverse Events were collected and assessed during each study visit during the 12 week treatment period and 4 week follow-up period.
Arm/Group | Lidocaine/Diphenhydramine (Combination) | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/27
Other Adverse Events (participants affected / at risk) | 30/39 | 30/39 | 23/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lidocaine/Diphenhydramine (Combination) (N=39) | Lidocaine (N=39) | Placebo (N=27)
Nasopharyngitis (Infections and infestations) | 7 | 4 | 6
Fungal infection (Infections and infestations) | 3 | 4 | 2
Vaginal candidiasis (Infections and infestations) | 2 | 4 | 2
Urinary tract infection (Infections and infestations) | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 4 | 4
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 4 | 3 | 4
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 | 4 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 5 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0
Headache (Nervous system disorders) | 8 | 5 | 3
Pain (General disorders) | 3 | 0 | 2
Pyrexia (General disorders) | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Multiple allergies (Immune system disorders) | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued following enrollment of 106 of the planned 140 participants due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish, or seek to publish, either in whole or in part, any results of the Clinical Investigation without the written consent of the Sponsor.